CLINICAL TRIAL: NCT00563264
Title: KAN-DO: A Family-based Intervention to Prevent Childhood Obesity
Acronym: KAN-DO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00007666; DK075439-01; 8609 (Other: Duke legacy protocol number)
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2013-08

CONDITIONS: Obesity; Prevention & Control; Postpartum Period
Keywords: obesity; parenting; postpartum period; family research
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Participants receive monthly newsletter (for 10 months) including general health and reading information for child and mother and incentives for completing the baseline and 2 follow-up assessments
  Interventions: Behavioral: KAN-DO
- 2 (Experimental): Mothers and preschoolers in the intervention group will receive monthly mailed family kits that encourage interactive mother/child exercises for healthy lifestyle change. Mailings are supported by counseling calls and two in-person motivational/informational group sessions. The content of the intervention addresses parenting skills, healthy eating, and physical activity. Families can earn $40 for returning postcards describing their activities in the past month.
  Interventions: Behavioral: KAN-DO

INTERVENTIONS:
Behavioral: KAN-DO — The 10 month KAN-DO intervention includes eight mailed interactive activity modules involving both the preschooler and mother that include relevant printed materials emphasizing parenting skills, healthy eating habits and increased physical activity. Mailed kits will each be followed by a supportive telephone counseling session based on motivational interviewing techniques. Mailed modules and telephone calls will be supplemented with two in-person motivational and informational sessions (at the beginning and in the middle of the intervention period).
  The Active Comparator group will receive monthly newsletters over the 10 month period related to boosting reading skills in their preschool children.

SUMMARY:
The purpose of this study is to evaluate the efficacy of an intervention (KAN-DO: Kids & Adults Now - Defeat Obesity) encouraging postpartum mothers and their preschool-aged children to work together to promote healthy eating, increase physical activity, and reduce sedentary behaviors. Via instruction in parenting skills and behavior change strategies, the goal is relative weight maintenance in children of healthy weight, and relative weight reduction in overweight children. The intervention will focus on a child (2-5 years of age) and his or her overweight or obese mother, who has just delivered a second or subsequent baby.

DETAILED DESCRIPTION:
OVERVIEW

The purpose of the study is to evaluate the efficacy of an intervention encouraging postpartum mothers and their preschool-aged children to work together to promote healthy eating, increase physical activity, and reduce sedentary behaviors. Via instruction in parenting skills and behavior change strategies, the end goal is relative weight maintenance in children of healthy weight, and relative weight reduction in overweight children. The intervention will focus on a preschooler (2-5 years of age) and his or her overweight or obese mother, who has just delivered a second or subsequent baby. 400 mother/preschooler dyads from the Triad and Triangle areas of NC will be randomized to:

THE CONTROL ARM Mothers in the control arm will receive a monthly newsletter, and be given monetary incentives to complete the baseline and follow-up assessments; or

THE KAN-DO INTERVENTION ARM Mothers and preschoolers in the intervention group will receive monthly mailed family kits that encourage interactive mother/child exercises for healthy lifestyle change. Mailings are supported by counseling calls and two in-person motivational/informational group sessions. The content of the intervention addresses parenting skills, healthy eating, and physical activity. Families can earn $40 for returning postcards describing their activities in the past month.

PRIMARY AIMS of the study address weight and behavior change in the child. SECONDARY AIMS of the study address expected healthy changes in the mother. Further, we will investigate the roles of parenting skills.

RECRUITMENT Eligible households contain a woman with a current postpartum BMI > 25 who has delivered a child in the past 6 months, and who has another child between the ages of 2 and 5.

SCREENING AND ELIGIBILITY:

At ~6 weeks postpartum, all women will be contacted by study staff and will have the study fully described. If women are interested, they will complete a brief set of questions to assess eligibility criteria, including: recent delivery of a baby, a preschooler in the home (2-5 years old), and a current BMI ≥25 (a confirmatory BMI ≥25 measured at baseline will be required for final inclusion). As part of the screening interview, women will also be asked questions to determine if either mother or preschooler has any conditions that would exclude them medically from the study. Eligible and interested families will be told that their family will be assigned at random to one of the research groups.

CONSENT:

Mother/child dyads that are deemed eligible and are willing to participate will attend a personal consent and baseline data collection appointment either at the Duke or UNC-G site. Women will bring their 2-5 year old child to this appointment. Consenting families will complete a survey, be weighed and measured, wear an activity monitor for a week and complete a dietary recall over the phone.

FOLLOW-UP Mother/child dyads will be contacted again at 12 and 24 months postpartum for final assessments. The 12 assessments are similar in scope to the baseline visit.

ELIGIBILITY:
Inclusion Criteria:

* Recent delivery of a baby (~6 months ago)
* A preschooler in the home (2-5 years old), and a current BMI ≥25 (with confirmatory BMI ≥25 measured at baseline
* Knowledge of English
* Regular access to a telephone and mailing address
* Mother's age of 18 or older
* Willingness to participate in a healthy lifestyle correspondence and telephone intervention.

Exclusion Criteria:

* Not meeting inclusion criteria
* Medical conditions preventing mother from walking a mile without assistance
* Conditions preventing the child from regular activity

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 832 (Actual)
Dates: Start 2007-10; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
BMI z-score (via measured weight and height) of preschooler | ~2 years post baseline

SECONDARY OUTCOMES:
Mother's measured weight, as well as eating and physical activity behavioral targets (brief measures) in both mother and child | ~12 and ~24 months post baseline

CONTACTS AND LOCATIONS:
Overall Officials: Truls Ostbye, MD PhD, Principal Investigator — Duke University; Cheryl Lovelady, PhD, RD, Principal Investigator — University of North Carolina, Greensboro
Locations (2):
- United States (2):
  - Duke University Dept. of Community and Family Medicine, Durham, North Carolina
  - UNC Greensboro, Greensboro, North Carolina

REFERENCES:
- [Background] Ostbye T, Zucker NL, Krause KM, Lovelady CA, Evenson KR, Peterson BL, Bastian LA, Swamy GK, West DG, Brouwer RJ. Kids and adults now! Defeat Obesity (KAN-DO): rationale, design and baseline characteristics. Contemp Clin Trials. 2011 May;32(3):461-9. doi: 10.1016/j.cct.2011.01.017. Epub 2011 Feb 18. PMID 21300177
- [Background] Dolinsky DH, Brouwer RJ, Evenson KR, Siega-Riz AM, Ostbye T. Correlates of sedentary time and physical activity among preschool-aged children. Prev Chronic Dis. 2011 Nov;8(6):A131. Epub 2011 Oct 17. PMID 22005624
- [Background] Wiltheiss GA, Lovelady CA, West DG, Brouwer RJ, Krause KM, Ostbye T. Diet quality and weight change among overweight and obese postpartum women enrolled in a behavioral intervention program. J Acad Nutr Diet. 2013 Jan;113(1):54-62. doi: 10.1016/j.jand.2012.08.012. Epub 2012 Nov 10. PMID 23146549
- [Result] Ostbye T, Krause KM, Stroo M, Lovelady CA, Evenson KR, Peterson BL, Bastian LA, Swamy GK, West DG, Brouwer RJ, Zucker NL. Parent-focused change to prevent obesity in preschoolers: results from the KAN-DO study. Prev Med. 2012 Sep;55(3):188-95. doi: 10.1016/j.ypmed.2012.06.005. Epub 2012 Jun 13. PMID 22705016
- [Derived] Ostbye T, Malhotra R, Stroo M, Lovelady C, Brouwer R, Zucker N, Fuemmeler B. The effect of the home environment on physical activity and dietary intake in preschool children. Int J Obes (Lond). 2013 Oct;37(10):1314-21. doi: 10.1038/ijo.2013.76. Epub 2013 May 20. PMID 23736357